CLINICAL TRIAL: NCT06548269
Title: Multimodal Prognostic Assessment of Acute Ischemic Stroke Patients With Atrial Fibrillation: a Prospective, Multicenter, Observational Study (IAT-CLOSURE)
Status: Recruiting | Type: Observational
Sponsor: Jinan Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IAT-CLOSURE
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-12

CONDITIONS: Acute Ischemic Stroke; Atrial Fibrillation
Keywords: Acute Ischemic Stroke; Atrial fibrillation; AF burden; Left atrial appendage closure
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with acute ischemic stroke and atrial fibrillation: Adult patients with an acute ischemic stroke and atrial fibrillation will undergo a baseline work-up and cardiologic work-up. Baseline work-up includes admission 12-lead ECG，blood analysis, brain CT/MRI, brain CTA/MRA/vessel ultrasound. Cardiologic work-up includes prolonged ECG monitoring, echocardiography and cardiac CTA. Treatment will follow the current guidelines.
  Interventions: Diagnostic Test: Cardiologic work-up

INTERVENTIONS:
Diagnostic Test: Cardiologic work-up — Noninvasive prolonged ECG monitoring with a duration of 7 days measuring AF burden； Echocardiography measuring LA volume or volume index, LA diameter or diameter index； Cardiac CTA measuring LAA morphologies, cardiac thrombus.

SUMMARY:
The main purpose of this study is to investigate the safety and outcomes of different treatment strategies, including best medical therapy (OAC [oral anticoagulation], antiplatelet [APT]) and left atrial appendage closure [LAAC] in acute ischemic stroke (AIS) patients with atrial fibrillation (AF) based on multimodal assessment from combined brain and cardiologic work-up, and to optimize secondary prevention.

DETAILED DESCRIPTION:
Ischemic stroke is the leading cause of disability and mortality globally. Atrial fibrillation（AF） is a well-established risk factor for ischemic stroke and responsible for up to one-third of all strokes. AF-related ischemic strokes are more frequently fatal or disabling than non-AF strokes. The overall prevalence of known or newly diagnosed AF in stroke patients is approximately 39.0%. Detecting underlying AF remains important for secondary prevention of recurrent stroke, with a different strategy from atherosclerotic cause of stroke. The increasingly common use of prolonged cardiac monitoring (PCM) after ischemic stroke has greatly increased the detection rates of previously undiagnosed AF in ischemic strokes, which was demonstrated by a series of trials. Additionally, AF burden, defined as percentage of the time in AF during cardiac monitoring, has been regarded as an important prognostic risk factor for thromboembolism.

Currently, the CHA2DS2-VASc score is the most widely used scoring system for assessing ischemic stroke risk in patients with AF and basis for initiation of anticoagulation. Anticoagulation is currently recommended for male with CHA2DS2-VASc score≥2 or female with CHA2DS2-VASc score≥3. Direct oral anticoagulants (DOACs) have been increasingly used in the past decade due to their similar to superior efficacy to vitamin K antagonists (VKAs), but a lower intracerebral bleeding risk in non-valvular atrial fibrillation (NVAF), defined as AF in the absence of moderate to severe mitral stenosis or a mechanical heart valve. For patients with AF who cannot tolerate long-term OACs due to various relative or absolute contraindications, left atrial appendage closure (LAAC) offers an alternative treatment strategy for these patients. Moreover, as one-third of patients with ischemic stroke and AF may have concomitant large artery atherosclerosis or small vessel disease, it is still unclear whether these patients should be left untreated or treated with antiplatelet (APT), DOACs, or with LAAC.

Traditional clinical practice mainly focuses on the presence of AF but rarely incorporates AF burden into a risk stratification scoring system. To our knowledge, no studies to date have investigated recurrent stroke risk stratification in AIS patients with AF based on AF burden assessed by PCM, not to mention guidance of treatment strategy selection. Further, other multimodal assessments, such as cerebral CT/MRI (e.g. infarct size and location), serum biomarkers (e.g. BNP, troponin, D-dimer levels) and cardiac structural markers (e.g. LA volume or volume index, LAA morphologies) have been reported as promising prognostic factors of stroke severity and recurrence. A comprehensive evaluation system is still lacking. In this prospective and multicenter registry study, we determine to test the safety and effectiveness of best medical therapy (OAC, APT) and LAAC using multimodal assessment from combined brain and cardiologic work-up, with the aim to optimize secondary prevention in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old；
2. Acute ischemic stroke with onset ≤ 14 days；
3. Previously or during this hospitalization diagnosed with non-valvular atrial fibrillation;
4. Informed consent obtained from the patient or his/her legal representative；

Exclusion Criteria:

1. Pacemaker, implantable cardioverter defibrillator or implantable cardiac monitor;
2. Left atrial appendage has been removed or post occlusion device implantation;
3. Transient AF secondary to other reversible disorders；
4. Life expectancy less than 1 year;
5. Patients that cannot complete subsequent follow-up (e.g. no fixed residence, overseas patients, etc.);
6. Females who are pregnant or in lactation;
7. Participating in other clinical trials that could confound the evaluation of the study;
8. Other circumstances that the investigator considers inappropriate for participation or may pose a significant risk to patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who had acute ischemic stroke symptoms within 7 days and previously or during this hospitalization diagnosed with non-valvular atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Composite endpoints of ischemic stroke, systemic embolism, myocardial infarction, major bleeding (BARC type 3-5) and all-cause mortality | 1 year
  Stroke only including ischemic stroke

SECONDARY OUTCOMES:
Composite endpoints of stroke, systemic embolism, myocardial infarction, major bleeding (BARC type 3-5) and all-cause mortality | 3 years
  Stroke including ischemic or hemorrhagic stroke

OTHER OUTCOMES:
Ischemic stroke | 12, 36months
  Rapid onset of a new focal neurological deficit with clinical and imaging evidence of infarction and not attributable to a non-ischemic etiology.
Hemorrhagic stroke | 12, 36months
  Hemorrhagic stroke is defined as an acute episode of focal or global cerebral or spinal dysfunction caused by a nontraumatic intraparenchymal, intraventricular, or subarachnoid hemorrhage
Systemic embolism | 12, 36months
  Systemic embolism was defined as an acute vascular occlusion of an extremity or organ confirmed by imaging or either surgery or autopsy.
Myocardial infarction (MI) | 12, 36months
  Myocardial infarction will be assessed according to the third universal definition of myocardial infarction (Eur Heart J, 2012).
BARC type 2 or 5 bleeding events | 12, 36months
  According to the BARC (Bleeding Academic Research Consortium) definition for bleeding
All-cause mortality | 12, 36months
  The occurrence of death from any cause
Changes in functional status based on Modified Rankin Scale | 12, 36months
  The Modified Rankin scale is used to measure the degree of disability or dependence in daily activities caused by a stroke. The scale runs from 0 to 6, from no symptoms (0) to death (6).
Changes in Barthel Index | 12, 36months
  The Barthel Index for Activities of Daily Living is uesd to measure a person's ability to complete activities of daily living (ADL).The total score range from 0 to 100, with higher scores indicating greater independence.
Relationship between atrial fibrillation burden and recurrent ischemic stroke | 12, 36months
  The association between atrial fibrillation burden measured from 7-day single lead ECG recorders and recurrent ischemic stroke
Complications related to left atrial appendage closure | within 12 months after surgery
  These complications may include pericardial effusion, device - related thrombosis, occluder detachment, stroke, and bleeding events.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinan Central Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No